CLINICAL TRIAL: NCT01126827
Title: Mindfulness-Based Cognitive Behavior Therapy for Bipolar Disorder: A Randomized, Controlled Study
Brief Title: Mindfulness-Based Cognitive Behavior Therapy for Bipolar Disorder
Acronym: MBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Thilo Deckersbach, PhD/Assistant Professor of Psychology, Harvard Medical School; Director, Cognitive Neuroscience Research, Bipolar Clinic and Research Program, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBCT Randomized Study
Record Dates: First submitted 2010-04-30; First posted 2010-05-20 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Mood Disorders; Residual Symptoms; Depression; Mania; Hypomania; Bipolar; Bipolar I; Bipolar II
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression; Mania

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supportive Psychotherapy (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Cognitive Behavioral Therapy or Supportive Psychotherapy
- Mindfulness-Based Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Cognitive Behavioral Therapy or Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Behavioral Therapy or Supportive Psychotherapy — 12 weekly group therapy sessions

SUMMARY:
The purpose of the study is to investigate the efficacy of mindfulness-based cognitive-behavior therapy (MBCT) for improvement of symptoms associated with bipolar disorder, by comparing MBCT to supportive psychotherapy. Patients who participate in this study will be randomly assigned to receive either

1. state of the art group MBCT, or
2. supportive group psychotherapy (which is considered part of the standard care available to patients at MGH).

DETAILED DESCRIPTION:
We will conduct a randomized controlled trial of group MBCT (n=30) vs. SP (n=30) and compare the benefits and durability of MBCT vs. SP for decreasing symptoms in DSM-IV bipolar individuals over a 12-week period adjunctive to mood stabilizing medications coupled with individual-therapy sessions. We will also conduct follow-up assessments at 3, 6, 9, and 12 months after the active phase of the study. Subjects in the MBCT group will receive group therapy sessions of standardized yoga-meditation based exercises enhanced by psychoeducation and relapse prevention for bipolar disorder. Subjects in the SP group will receive support for coping with the symptoms of bipolar disorder, as well as psychoeducation about bipolar disorder. The focus of SP is on reflecting and expressing feelings about current life issues. Patients are supported and comforted when coping with difficult situations, depression, mood swings, or anger. We will assess mood, cognitive and psychosocial functioning before and after treatment for participants in both groups. Finally, we will investigate the functional neuroanatomy associated with memory impairment, attention, and mindful breathing in subjects with bipolar disorder as a predictor of treatment response using functional Magnetic Resonance Imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* MINI diagnostic criteria for any bipolar disorder (type I, type II, and NOS)
* Written informed consent
* Men or women aged 18-65
* No episodes of mania in the previous 4 weeks.
* Able to read and understand English.

Exclusion Criteria:

* Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment.
* History of seizure disorder, brain injury, any history of known neurological disease (multiple sclerosis, degenerative disease such as ALS, Parkinson disease and any movement disorders, etc).
* History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, major depressive disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, including alcohol, active within the last 12 months.
* Patients who have untreated hypothyroidism.
* Patients who have had electroconvulsive therapy (ECT) within the 6 months preceding enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) & Young Mania Rating Scale (YMRS) | 12 weeks
  HAM-D (depression severity) and YMRS (mania/hypomania severity) total scores will be evaluated as the primary outcome measures of mood symptoms of bipolar disorder as part of this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Deckersbach, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Bipolar Clinic and Research Program, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hanssen I, Huijbers M, Regeer E, Lochmann van Bennekom M, Stevens A, van Dijk P, Boere E, Havermans R, Hoenders R, Kupka R, Speckens AE. Mindfulness-based cognitive therapy v. treatment as usual in people with bipolar disorder: A multicentre, randomised controlled trial. Psychol Med. 2023 Oct;53(14):6678-6690. doi: 10.1017/S0033291723000090. Epub 2023 Mar 7. PMID 39625263
- See also: MGH Bipolar Clinic and Research Program — http://www.massgeneral.org/bipolar